CLINICAL TRIAL: NCT05699343
Title: Surgical Treatment of Peri-implantitis Using a Bone Substitute With or Without a Resorbable Collagen Membrane. A Randomized Clinical Trial
Brief Title: Surgical Treatment of Peri-implantitis Using a Bone Substitute With or Without a Resorbable Collagen Membrane
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Ravida (Other)
Collaborators: SigmaGraft Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Andrea Ravida, Periodontics Program Director, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY22080031
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Peri-Implantitis; Surgery
Keywords: peri-implantitis; bone augmentation; collagen membrane; surgical treatment; dental implant
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: The present study will be a parallel, randomized single center clinical trial where participants will be randomized in to 2 groups: treatment with or without resorbable collagen membrane.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bone grafting with collagen membrane (Experimental): This arm will receive surgical intervention involving placement of a bone xenograft subsitute (InterOss Collagen) into the peri-implant bone defect with a collagen membrane (InterCollagen Guide) placed over the bone graft.
  Interventions: Procedure: InterOss Collagen (Bone xenograft) and InterOss Collagen Guide (Collagen membrane)
- Bone grafting without collagen membrane (Active Comparator): This arm will receive surgical intervention involving placement of a bone xenograft subsitute (InterOss Collagen) into the peri-implant bone defect with no collagen membrane placed over the graft.
  Interventions: Procedure: InterOss Collagen (Bone xenograft)

INTERVENTIONS:
Procedure: InterOss Collagen (Bone xenograft) and InterOss Collagen Guide (Collagen membrane) — Group will receive InterOss Collagen and InterOss Collagen Guide during surgical intervention visit.
  Arms: Bone grafting with collagen membrane
Procedure: InterOss Collagen (Bone xenograft) — Group will only receive InterOss Collagen during surgical intervention visit.
  Arms: Bone grafting without collagen membrane

SUMMARY:
The objective of the present randomized clinical trial will be to compare two surgical methods of treating peri-implantitis. This study will determine if surgical debridement of peri-implantitis bone defects, including air powder abrasive (APA) decontamination of implant surfaces, in combination with the placement of a bone graft, differs in treatment outcomes compared to placing the same bone graft material with a resorbable collagen membrane placed over the bone graft.

DETAILED DESCRIPTION:
The purpose of the study is to compare treatment outcomes of peri-implantitis defects when using a defect fill substitute (InterOss Collagen), against the treatment outcome when placing the same defect fill substitute with a resorbable collagen membrane (InterCollagen Guide). There is no current literature to suggest that placing a collagen membrane over a bone grafting material in an infrabony defect of more than 270 degrees is more effective than placing the bone graft material alone. The present study will help in understanding if such defects require an additional placement of a collagen membrane which could increase the cost of the procedure for the practitioner and the patient.

The study will be conducted at the University of Pittsburgh School of Dental Medicine Graduate Periodontics Department. A detailed description of research activities during each patient visit is provided below.

Screening Visit (V0):

Prior to starting any of the procedures, the subject will complete the informed consent interview. Patients will be screened to assess for inclusion in the study. Vitals (blood pressure and heart rate) will be measured and medical history will be discussed. Limited field of view (FOV) cone beam computed tomography (CBCT) scan will be taken and examined prior to the study to determine the presence of a 270 degree circumferential boney defect for inclusion in the study. Probing pocket depths (PPD), plaque sites, mobility and bleeding on probing (BOP) are clinical measurements that will be completed. The visit will take approximately 1.5 hours. All procedures will be performed by the faculty and Periodontics graduate resident.

Pre-surgical phase (V1):

If the patient is eligible and willing to participate in the study following the screening visit, they will return for V1. Their medical history will be reviewed, blood pressure and heart rate will be measured. Any adverse events from the previous visit will be assessed. A periapical (PA) radiograph will be taken to confirm a crater like defect >=3mm. The prosthetic superstructures (implant crowns) will be removed followed by placement of cover screws. PPD will be measured twice (with and without the implant crown). Bleeding on Probing (BOP), suppuration, mobility, and plaque sites will be recorded. Clinical photographs will be taken of the teeth and inside of the mouth. Generalized supragingival debridement will be performed. Patients will be informed that newly fabricated crowns might be needed after the treatment as part of the study. During this visit, patients will be also re-instructed and emphasized on maintaining proper at-home oral hygiene measures with a soft-bristled toothbrush for minimizing trauma to marginal soft tissues. The visit will take approximately 2 hours. All procedures will be performed by the faculty and Periodontics graduate resident.

Surgical treatment procedures (V2) After 4 to 6 weeks, the patient will undergo regenerative surgical procedure. Their medical history will be reviewed, blood pressure and heart rate will be measured. Any adverse events since the previous visit will be assessed. The Study individuals will receive a local anesthetic as needed by the surgeon. Intra-sulcular, and if necessary, vertical releasing incisions will be made. Soft tissue flaps will be elevated at buccal and lingual aspects providing adequate access. Granulation tissue and mineralized deposits at implants will be removed using titanium curettes. The implant surfaces will be decontaminated with airflow. Once the surgical site was debrided, clinical intra-surgical measurements will be made. The measurement of peri-implant defect depth will be made clinically intra-surgically. Defects will be measured by calibrated examiners using a periodontal probe. The depth will be measured to the deepest point of the defect. This will be termed the clinical vertical defect fill (DF), and assessed at each implant site (buccal, lingual/palatal, mesial, distal) as follows: DF = (Measurement at the surgical treatment) - (Measurement at re-entry procedure). The defect resolution (DR) on the other hand will be measured as the percentage of the defect that was filled with bone at the follow up compared to the original defect depth. The horizontal defect, width of keratinized tissue, and soft tissue thickness will also be measured at this visit.

Thereafter, study individuals will be randomized to control or test groups using the SPSS randomization method (SPSS PASW 23.0 statistical software package, SPSS Inc., Armonk, NY, USA). Depending on the randomization, one of the following therapies was used: (a) (control group); bone grafting alone (InterOss Collagen) will be placed. (b) (test group); the intraosseous component will be filled with bone grafting (InterOss Collagen) and covered with a resorbable collagen membrane (InterCollagen Guide). InterOss Collagen is an FDA cleared for use in guided bone regenerative procedures. InterOss Collagen is a bovine derived anorganic hydroxyapatite collagen composite composed of 90% bovine granules and 10% collagen fibers molded in a block form. InterCollagen Guide is an FDA cleared porcine derived resorbable collagen membrane intended for periodontal and dental surgeries. In both groups, if needed, a periosteal releasing incision will be made to allow complete coverage of the wound area. In both study groups, surgical soft tissue flaps will be sutured with interrupted sutures without tissue tension using 4/0 or 5/0 PGA providing full wound closure. Clinical photographs will be taken again, and surgical video may be recorded when possible. All study individuals will receive postoperative antibiotics and prescribed post-operative pain relievers, as well as care instructions.

The postoperative medications may include:

Amoxicillin 500 mg 3 x 7 days

* Clindamycin 300 mg 4 x 7 days Ibuprofen 600 mg PRN Chlorhexidine 0.12% rinse 2 x 2 weeks Tylenol 3 (300mg-30mg)* Medrol Dose Pack (as needed) Instructions not to wear any removable prosthesis during the healing phase
* Administer if drug allergy to Amoxicillin *Administer as alternative to Ibuprofen

The visit will take approximately 2.5-3 hours. All procedures will be performed by the faculty and Periodontics graduate resident.

4 weeks post op (V3) After 4 weeks (± 2 days), the patient will return for follow-up. Any changes to their medical history will be reviewed, blood pressure and heart rate will be measured. Any adverse events since the previous visit will be assessed. Sutures will be removed. Clinical photographs will be taken again. The visit will take approximately 0.5-1 hours. All procedures will be performed by the faculty and Periodontics graduate resident.

Re-entry procedure and replacement of superstructures (healing abutment) (V4) After 4 months of uninterrupted healing, patients will return for the re-entry procedure. Any changes to their medical history will be reviewed, blood pressure and heart rate will be measured. Any adverse events since the previous visit will be assessed. A standardized PA radiograph will be taken at this visit. Intrasulcular incision will be performed on the adjacent teeth and midcrestal incision at the implant location. Full thickness flap will be elevated, and the same defect measurements taken during the surgical procedures will be performed to obtain clinical changes in peri-implant bone levels. Where the defect fill will be measured as the difference in millimeters between the initial measurements taken at baseline and the depth of defect present at follow up. During the re-entry procedure, if the bone defect around the implant is not completely filled after V2, (it happens that we succeed to feel 60-70% of the defect, but not the whole defect), additional bone grafting material will be added after taking intra-surgical measurements. Please note the same bone graft material will be used, and will not involve additional clinical procedures, since the flap is open for the re-entry procedures. The outcome of "complete bone fill?" Yes/No will be recorded on the Visit form. Then, implant cover screws will be replaced by appropriate healing abutments, followed by single interrupted sutures for re-adaptation of the flap. Clinical photographs will be taken again, and surgical video may be recorded. Finally, a periodontal maintenance will be performed. The visit will take approximately 2 hours. All procedures will be performed by the faculty and Periodontics graduate resident. During this period, if needed new crowns will be designed, fabricated, and delivered to all patients and for all treated implants.

Post op after stage 2 (V5) Approximately 2 weeks after V4, subjects will return for V5. Any changes to their medical history will be reviewed, blood pressure and heart rate will be measured. Any adverse events since the previous visit will be assessed. Sutures will be removed. If a new crown is needed, digital impression will be taken with the Trios hand-held scanner, and patient will be referred to receive a new crown. If no new crown is needed, the old crown will be replaced at the next visit. Clinical photographs will be taken again. The visit will take approximately 1-2 hours. All procedures will be performed by the faculty and Periodontics graduate resident.

Crown placement/replacement (V6) Approximately 1 month after V5, the subjects will return for the Implant Crown replacement. Any changes to their medical history will be reviewed, blood pressure and heart rate will be measured. Any adverse events since the previous visit will be assessed. The old crown or the new crown will be placed in the treated area. A radiograph may be taken to assist in placement. The visit will take approximately 1- 2 hours. All procedures will be performed by the faculty and Periodontics graduate resident.

8 months visit (V7) For V7, subjects will return at approximately 8-months post-op. Any changes to their medical history will be reviewed, blood pressure and heart rate will be measured. Any adverse events since the previous visit will be assessed. Probing pocket depth (PPD), recession, BOP, plaque, suppuration and mobility measurement will be recorded. Radiographic measurements (bone fill) will be obtained as performed at the pre-surgical visit (time point 1). Dental prophylaxis and periodontal maintenance will be performed. Clinical photographs will be taken again. The visit will take approximately 0.5-1 hours. All procedures will be performed by the faculty and Periodontics graduate resident.

12 months visit (V8) Any changes to subject's medical history will be reviewed, blood pressure and heart rate will be measured. Any adverse events since the previous visit will be assessed. Probing pocket depth (PPD), recession, BOP, suppuration, mobility and plaque measurements will be taken as in previous visits. Radiographic measurements (bone fill) will be obtained as performed at the pre-surgical visit (time point 1) using a standardized PA radiograph. Periodontal maintenance will be performed. Clinical photographs will be taken again. The visit will take approximately 0.5-1 hours. All procedures will be performed by the faculty and Periodontics graduate resident.

Year 2:

15, 18, 21, 24 months visit (V9, V10, V11, V12) Any changes to subject's medical history will be reviewed, blood pressure and heart rate will be measured. Any adverse events since the previous visits will be assessed. Probing pocket depth (PPD), recession, BOP, suppuration, mobility and plaque measurements will be taken as in previous visits. Radiographic measurements (bone fill) will be obtained as performed at the last visit (V12, timepoint 24 months) using a standardized PA radiograph. If a patient is pregnant, the periapical x-ray will not be performed. Periodontal maintenance will be performed. Clinical photographs will be taken again. The visit will take approximately 0.5-1 hours. All procedures will be performed by the faculty and Periodontics graduate resident.

Year 3:

27, 30, 33, 36 months visit (V13, V14, V15, V16) Any changes to subject's medical history will be reviewed, blood pressure and heart rate will be measured. Any adverse events since the previous visits will be assessed. Probing pocket depth (PPD), recession, BOP, suppuration, mobility and plaque measurements will be taken as in previous visits. Radiographic measurements (bone fill) will be obtained as performed at the last visit (V16, timepoint 36 months) using a standardized PA radiograph. If a patient is pregnant, the periapical x-ray will not be performed. Periodontal maintenance will be performed. Clinical photographs will be taken again. The visit will take approximately 0.5-1 hours. All procedures will be performed by the faculty and Periodontics graduate resident.

Year 4:

39, 42, 45, 48 months visit (V17, V18, V19, V20) Any changes to subject's medical history will be reviewed, blood pressure and heart rate will be measured. Any adverse events since the previous visits will be assessed. Probing pocket depth (PPD), recession, BOP, suppuration, mobility and plaque measurements will be taken as in previous visits. Radiographic measurements (bone fill) will be obtained as performed at the last visit (V20, timepoint 48 months) using a standardized PA radiograph. If a patient is pregnant, the periapical x-ray will not be performed. Periodontal maintenance will be performed. Clinical photographs will be taken again. The visit will take approximately 0.5-1 hours. All procedures will be performed by the faculty and Periodontics graduate resident.

Year 5:

51, 54, 57, 60 months visit (V21, V22, V23, V24) Any changes to subject's medical history will be reviewed, blood pressure and heart rate will be measured. Any adverse events since the previous visits will be assessed. Probing pocket depth (PPD), recession, BOP, suppuration, mobility and plaque measurements will be taken as in previous visits. Radiographic measurements (bone fill) will be obtained as performed at the last visit (V24, timepoint 60 months) using a standardized PA radiograph. If a patient is pregnant, the periapical x-ray will not be performed. Periodontal maintenance will be performed. Clinical photographs will be taken again. The visit will take approximately 0.5-1 hours. All procedures will be performed by the faculty and Periodontics graduate resident.

Clinical measurements:

* The following baseline procedures will be performed; (a) Intra-oral photographs and intra-oral radiographs of the implant sites; (b) clinical recording of full mouth plaque scores (FMPS) (presence of dental plaque along the peri-implant mucosal margin (gingival margin at teeth) was expressed as a percentage of examined sites within each subject including four sites per tooth and implant, (c) clinical recording of local plaque score (LPS) (presence of dental plaque along the mucosal margin at four sites of each treated implant and expressed as a percentage of implant sites within each subject), (d) clinical recording of probing pocket depths (PPD) (at all teeth, and the specific implant in the study (four sites; implant/tooth) to the nearest millimeter with a North Carolina probe (e) clinical recording of full mouth bleeding scores calculated as the percentage of assessed surfaces with BOP, (f) BOP will also be assessed with the North Carolina probe at four sites per implant. The bleeding will be graded; 0 = no bleeding, 1 = dot of bleeding, 2 = line of bleeding and 3 = drop of bleeding (Mombelli, van Oosten, Schurch, & Lang, 1987), (g) clinical recording of recession at the peri-implant mucosal margin (buccal/lingual-palatal) relative to a fixed reference point on implants and (h), clinical recording of presence/absence of suppuration (SUP) at the implant (4 sites/implant).
* Peri-implant defect depth will be made clinically intra-surgically. Defects will be measured by calibrated examiners using a periodontal probe. The depth will be measured to the deepest point of the defect. This will be termed the clinical vertical defect fill (DF), and assessed at each implant site (buccal, lingual/palatal, mesial, distal) as follows: DF = (Measurement at the surgical treatment) - (Measurement at re-entry procedure). The defect resolution (DR) will be measured as the percentage of the defect that was filled with bone at the follow up compared to the original defect depth.
* MBL will be calculated based on standardized radiographs using registered bite-block with a Rinn (Dentsply Rinn, Elgin, IL, USA) film holder and expressed as the distance from the implant shoulder to the most coronal bone-to-implant contact (BIC) on the mesial and distal side of the implant. The mean values will be calculated for each implant. In the case that the bone levels around the study implants are hidden or difficult to read, new radiographs will be taken. Peri-implant marginal bone levels will be measured using the ImageJ software* (ImageJ, U. S. National Institutes of Health, Bethesda, Maryland, USA) (Schneider, Rasband, & Eliceiri, 2012). The software will be calibrated for every single image using the known implant length or the length of the implant collar. Measurements of the mesial and distal bone crest level adjacent to each implant will be rounded to the nearest 0.1 mm. Implants with bone up to the coronal margin of the implant collar will be given a value of zero. Mesial and distal measurements of each implant are averaged, and a mean calculated at patient level and then at group level. Implant failure: It will be defined as implant mobility (assessed from force applied with two hand instrument), pain, or neuropathy. Composite definition of successful treatment outcome: A composite therapeutic endpoint composed of no evidence of BOP or evidence of BOP grade 1 and with no suppuration at any of four assessed sites per implant PPD ≤5 mm, and with ≥1.0 mm defect fill will be used to define a successful treatment outcome. Thickness of soft tissues will be measured with a 1.0-mm marked periodontal probe (UNC, Hu-Friedy, Chicago, IL, USA) on the top of bone crest in the center of the implant. This will ensure direct visibility of mucosal thickness during measurement.

ELIGIBILITY:
Inclusion Criteria: To be enrolled, the participant must meet the following inclusion criteria:

1. age 18 years or older
2. be patients of record at the University of Pittsburgh Periodontics Department
3. Systemically healthy patients
4. Full-mouth plaque score and full-mouth bleeding score ≤ 30% (measured at six sites per tooth)
5. Study individuals will be included if they met the following criteria: (a) one or more peri-implant sites with PPD ≥6 mm combined with BOP/suppuration, and (b) peri-implant marginal bone loss, defined as a crater like defect ≥3 mm as assessed from intra- oral radiographs, (c) Infrabony circumferential defect of more than 270° determined by CBCT, (d) crown not possible to retrieve before surgery

Exclusion Criteria:study individuals will be excluded if any of the folllowing apply:

1. Unlikely to be able to comply with study procedures and unable to return to SDM for multiple appointments over the course of about a year.
2. Uncontrolled pathologic processes in the oral cavity (cancer and active periodontal disease)
3. History of allergic reactions to dental local anesthetics
4. History of head and neck chemotherapy or radiation within 5 years prior to surgery
5. Systemic or local disease or condition that could compromise post-operative healing and/or osseointegration, such as HIV infection, Paget's disease, osteoporosis, etc.
6. Reported diagnosis of diabetes mellitus
7. Patients taking corticosteroids, IV bisphosphonates, or any immunosuppressant medication that could influence post-operative healing and/or osseointegration
8. Smokes more than 10 cigarettes/day (self-reported)
9. History or current medications with known side effects of gingival growth (including any of the following: phenytoin, phenobarbital, lamotrigine, vigabatrin, ethosuximide, topiramate, primidone, nifedipine, diltazem, amlodipine, felodipine, verapamil, cyclosporine).
10. Present alcohol and/or drug abuser (self-reported)
11. Pregnant, unsure pregnancy status, or lactating females (self-reported), or planning to become pregnant within 1 year of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Successful Treatment of Peri-Implantitis | 1 year
  Composite definition of successful treatment outcome: A composite therapeutic endpoint composed of no evidence of BOP or evidence of BOP grade 1 and with no suppuration at any of four assessed sites per implant PPD ≤5 mm, and with ≥1.0 mm defect fill will be used to define a successful treatment outcome. Thickness of soft tissues will be measured with a 1.0 mm marked periodontal probe (UNC, Hu-Friedy, Chicago, IL, USA) on the top of bone crest in the center of the implant. This will ensure direct visibility of mucosal thickness during measurement.
  Definition of unsuccessful treatment will mean that the implant does not meet successful treatment outcome criteria or if an implant failure occurs. Implant failure will be defined as implant mobility (assessed from force applied with two hand instrument), pain, or neuropathy.
  These criteria will be assessed at 12 months post surgery. All subjects will be followed for 5 years and the same outcome will be assessed yearly.
Successful Treatment of Peri-Implantitis | 2 years
  Composite definition of successful treatment outcome: A composite therapeutic endpoint composed of no evidence of BOP or evidence of BOP grade 1 and with no suppuration at any of four assessed sites per implant PPD ≤5 mm, and with ≥1.0 mm defect fill will be used to define a successful treatment outcome. Thickness of soft tissues will be measured with a 1.0 mm marked periodontal probe (UNC, Hu-Friedy, Chicago, IL, USA) on the top of bone crest in the center of the implant. This will ensure direct visibility of mucosal thickness during measurement.
  Definition of unsuccessful treatment will mean that the implant does not meet successful treatment outcome criteria or if an implant failure occurs. Implant failure will be defined as implant mobility (assessed from force applied with two hand instrument), pain, or neuropathy.
  These criteria will be assessed at 24 months post surgery. All subjects will be followed for 5 years and the same outcome will be assessed yearly.
Successful Treatment of Peri-Implantitis | 3 years
  Composite definition of successful treatment outcome: A composite therapeutic endpoint composed of no evidence of BOP or evidence of BOP grade 1 and with no suppuration at any of four assessed sites per implant PPD ≤5 mm, and with ≥1.0 mm defect fill will be used to define a successful treatment outcome. Thickness of soft tissues will be measured with a 1.0 mm marked periodontal probe (UNC, Hu-Friedy, Chicago, IL, USA) on the top of bone crest in the center of the implant. This will ensure direct visibility of mucosal thickness during measurement.
  Definition of unsuccessful treatment will mean that the implant does not meet successful treatment outcome criteria or if an implant failure occurs. Implant failure will be defined as implant mobility (assessed from force applied with two hand instrument), pain, or neuropathy.
  These criteria will be assessed at 36 months post surgery. All subjects will be followed for 5 years and the same outcome will be assessed yearly.
Successful Treatment of Peri-Implantitis | 4 years
  Composite definition of successful treatment outcome: A composite therapeutic endpoint composed of no evidence of BOP or evidence of BOP grade 1 and with no suppuration at any of four assessed sites per implant PPD ≤5 mm, and with ≥1.0 mm defect fill will be used to define a successful treatment outcome. Thickness of soft tissues will be measured with a 1.0 mm marked periodontal probe (UNC, Hu-Friedy, Chicago, IL, USA) on the top of bone crest in the center of the implant. This will ensure direct visibility of mucosal thickness during measurement.
  Definition of unsuccessful treatment will mean that the implant does not meet successful treatment outcome criteria or if an implant failure occurs. Implant failure will be defined as implant mobility (assessed from force applied with two hand instrument), pain, or neuropathy.
  These criteria will be assessed at 48 months post surgery. All subjects will be followed for 5 years and the same outcome will be assessed yearly.
Successful Treatment of Peri-Implantitis | 5 years
  Composite definition of successful treatment outcome: A composite therapeutic endpoint composed of no evidence of BOP or evidence of BOP grade 1 and with no suppuration at any of four assessed sites per implant PPD ≤5 mm, and with ≥1.0 mm defect fill will be used to define a successful treatment outcome. Thickness of soft tissues will be measured with a 1.0 mm marked periodontal probe (UNC, Hu-Friedy, Chicago, IL, USA) on the top of bone crest in the center of the implant. This will ensure direct visibility of mucosal thickness during measurement.
  Definition of unsuccessful treatment will mean that the implant does not meet successful treatment outcome criteria or if an implant failure occurs. Implant failure will be defined as implant mobility (assessed from force applied with two hand instrument), pain, or neuropathy.
  These criteria will be assessed at 60 months post surgery. All subjects will be followed for 5 years and the same outcome will be assessed yearly.

SECONDARY OUTCOMES:
Radiographic Marginal Bone Loss (MBL) | 8 months
  Marginal bone loss (MBL) will be calculated based on standardized radiographs using registered bite-block with a film holder and expressed as the distance from the implant shoulder to the most coronal bone-to-implant contact (BIC) on the mesial and distal side of the implant. The mean values will be calculated for each implant. Peri-implant marginal bone levels will be measured using the ImageJ software. The software will be calibrated for every single image using the known implant length or the length of the implant collar. Measurements of the mesial and distal bone crest level adjacent to each implant will be rounded to the nearest 0.1 mm. Implants with bone up to the coronal margin of the implant collar will be given a value of zero. Mesial and distal measurements of each implant are averaged, and a mean calculated at patient level.
Radiographic Marginal Bone Loss (MBL) | 12 months
  MBL will be calculated based on standardized radiographs using registered bite-block with a film holder and expressed as the distance from the implant shoulder to the most coronal bone-to-implant contact (BIC) on the mesial and distal side of the implant. The mean values will be calculated for each implant. Peri-implant marginal bone levels will be measured using the ImageJ software. The software will be calibrated for every single image using the known implant length or the length of the implant collar. Measurements of the mesial and distal bone crest level adjacent to each implant will be rounded to the nearest 0.1 mm. Implants with bone up to the coronal margin of the implant collar will be given a value of zero. Mesial and distal measurements of each implant are averaged, and a mean calculated at patient level.
Peri-Implant Bleeding on Probing | 8 months
  Clinical measurements will be taken at 8 months following the surgical procedure and compared to baseline measurements. Following probing measurements, bleeding on probing will be recorded at 6 sites around the implant (mesial facial, distal facial, facial, mesial lingual, distal lingual and lingual). Bleeding will be recorded as present if bleeding occurs within 30 seconds of probing a site and will be recorded as absent if no bleeding occurs.
Peri-Implant Bleeding on Probing | 12 months
  Clinical measurements will be taken at 12 months following the surgical procedure and compared to baseline measurements. Following probing measurements, bleeding on probing will be recorded at 6 sites around the implant (mesial facial, distal facial, facial, mesial lingual, distal lingual and lingual). Bleeding will be recorded as present if bleeding occurs within 30 seconds of probing a site and will be recorded as absent if no bleeding occurs.
Peri-Implant Probing Depth | 8 months
  Clinical measurements will be taken at 8 months following the surgical procedure and compared to baseline measurements. Probing depths will be recorded on 6 sites around the implant (mesial facial, distal facial, facial, mesial lingual, distal lingual and lingual). All clinical measurements will be made in millimeters and measured using a standard periodontal probe and by one examiner.
Peri-Implant Probing Depth | 12 months
  Clinical measurements will be taken at 12 months following the surgical procedure and compared to baseline measurements. Probing depths will be recorded on 6 sites around the implant (mesial facial, distal facial, facial, mesial lingual, distal lingual and lingual). All clinical measurements will be made in millimeters and measured using a standard periodontal probe and by one examiner.
Clinical Peri-Implant Bone Defect Fill | 4 months
  Peri-implant bone defect depth will be measured clinically during initial surgical procedure and at uncovery to determine clinical bone defect fill (DF). The bone defect will be measured using a prefabricated acrylic stent stabilized on adjacent teeth. The depth will be measured from the marked area of the stent to the deepest point of the defect using a standard periodontal probe and recorded in mm. This will be termed the clinical vertical defect fill (DF), and assessed at each implant site (buccal, lingual/palatal, mesial, distal) as follows: DF = (Measurement at the surgical treatment) - (Measurement at re-entry procedure).
Clinical Peri-Implant Bone Defect Resolution | 4 months
  Peri-implant bone defect depth will be measured clinically during initial surgical procedure and at uncovery to determine bone defect resolution. The bone defect will be measured using a prefabricated acrylic stent stabilized on adjacent teeth. The depth will be measured from the marked area of the stent to the deepest point of the defect using a standard periodontal probe and recorded in mm. The defect resolution (DR) will be measured as the percentage of the defect that was filled with bone at the follow up compared to the original defect depth.
Patient Reported Pain Outcomes | 2 weeks
  Patients will be provided with numerical pain assessment forms following each surgical intervention and these forms will be collected at the post operative visits. Patients will be instructed to record post operative pain using a numerical Pain Scale with 0 being no pain and 10 being the worst pain. Patients will begin recording pain scales starting the day of surgery and continue daily for 7 days. Patient will return the completed form at the 2 week post operative visit following the uncovery surgical procedure. This data will be used to assess if there are any differences in patient reported pain outcomes between both groups.
Patient Reported Pain Outcomes | 4 weeks
  Patients will be provided with numerical pain assessment forms following each surgical intervention and these forms will be collected at the post operative visits. Patients will be instructed to record post operative pain using a numerical Pain Scale with 0 being no pain and 10 being the worst pain. Patients will begin recording pain scales starting the day of surgery and continue daily for 7 days. Patient will return the completed form at the 4 week post operative visit following the first surgical procedure. This data will be used to assess if there are any differences in patient reported pain outcomes between both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ravida, DDS MS PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Dental Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Research study data will be stored separately from medical records. Consent forms and copies of letters/correspondence will be stored separately from the research data. Data will be coded with a participant code number which will be assigned consecutively as subjects are enrolled. There will be an excel spreadsheet containing the linkage code to the identifiable patient name or Axium number. This spreadsheet will be password protected and only accessible to the research team and will be saved in a separate location then the medical records (such as OneDrive).
  De-identified research data will be shared with the sponsor and may be shared with other researchers studying similar conditions.
  In any publication of this data, confidentiality of individual subjects will be protected.
  De-identified data may be shared with other researchers or federal repositories in the future under an approved sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available at completion of study and be available for 7 years following final reporting.
Access Criteria: Access to identifiable information will only be granted to authorized representatives from the University of Pittsburgh's Office of Research Protections who may review information to monitor the conduct of this study.
  De-identified data will be shared with the study sponsor, Sigma Graft Inc. This de-identified information may also be used by other researchers for future research studies.